CLINICAL TRIAL: NCT00112723
Title: A Phase I/II Study of Flavopiridol Administered as a 30-Minute Bolus Followed by a 4-Hour Infusion in Lymphomas and Multiple Myeloma
Brief Title: Flavopiridol in Treating Patients With Relapsed or Refractory Lymphoma or Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Administratively Complete
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01346; NCI-2011-01346 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU-04100; CDR0000429577; OSU-2005C0006; NCI-7002; OSU 04100 (Other: Ohio State University Medical Center); 7002 (Other: CTEP); U01CA076576 (NIH); N01CM00070 (NIH); P30CA016058 (NIH)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-06

CONDITIONS: Adult Lymphocyte Depletion Hodgkin Lymphoma; Adult Lymphocyte Predominant Hodgkin Lymphoma; Adult Mixed Cellularity Hodgkin Lymphoma; Adult Nodular Sclerosis Hodgkin Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Multiple Myeloma; Splenic Marginal Zone Lymphoma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — alvocidib

ARMS (1):
- Treatment (alvocidib) (Experimental): PHASE I: Patients receive flavopiridol IV over 4½ hours on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  PHASE II: Patients receive flavopiridol* as in phase I at the MTD determined in phase I.
  Interventions: Drug: alvocidib

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275

SUMMARY:
This phase I/II trial is studying the side effects and best dose of flavopiridol and to see how well it works in treating patients with lymphoma or multiple myeloma. Drugs used in chemotherapy, such as flavopiridol, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the disease-specific dose-limiting toxicity and maximum tolerated dose of flavopiridol in patients with relapsed or refractory lymphoma or multiple myeloma.

II. Determine the complete and partial response rate in patients with selected non-Hodgkin's lymphoma (e.g., indolent B-cell, mantle cell, intermediate grade B-cell, and T/NK-cell), Hodgkin's lymphoma, or multiple myeloma treated with this drug.

III. Determine the qualitative and quantitative toxic effects or this drug, in terms of organ specificity, time course, predictability, and reversibility in these patients.

IV. Determine subsets of lymphoid/plasma cell malignancies that are suitable for larger phase II studies designed to further evaluate the efficacy and toxicity of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics of this drug in these patients. II. Determine the effect of this drug on innate immunity (including T-, B-, and NK-cell subsets) and quantitative immunoglobulin levels in these patients.

III. Determine whether acute infusion toxicity (e.g., fever, hypotension, tumor pain, and dyspnea) observed with other flavopiridol treatment schedules is related to a cytokine-release syndrome in these patients.

IV. Determine whether this drug induces response (independent of p53 mutational status) in these patients.

OUTLINE: This is a phase I, dose-escalation study followed by a multicenter, phase II, pilot study. Patients enrolled in the phase II portion of the study are stratified according to diagnosis.

PHASE I: Patients receive flavopiridol IV over 4½ hours on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PHASE II: Patients receive flavopiridol* as in phase I at the MTD determined in phase I.

NOTE: The phase II treatment dose and schedule for hairy cell leukemia patients will be adapted from that developed in previous phase II studies of flavopiridol for the treatment of chronic lymphocytic leukemia.

After completion of study therapy, patients are followed every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following hematologic malignancies:

  * Hodgkin's lymphoma
  * Non-Hodgkin's lymphoma (NHL)
  * Multiple myeloma
* Patients in the phase II portion of the study are enrolled in 1 of the following strata according to diagnosis*

  * Stratum 1: Indolent B-cell NHL (non-Hodgkin's lymphoma), follicle center B-cell NHL (grade 1, 2, or 3), marginal zone lymphoma, Waldenstrom's macroglobulinemia, or small lymphocytic lymphoma (without blood lymphocytosis at any point in the disease process)

    * Must have progressive lymphadenopathy, worsening cytopenias, or progressive symptoms attributed to lymphoma
    * Must require therapy, as determined by progressive anemia, thrombocytopenia, symptoms (e.g., fever, night sweats, weight loss, or fatigue), or progressive lymphadenopathy that causes discomfort
    * Received ≥ 2 prior therapies, including rituximab
  * Stratum 1a: Hairy cell leukemia

    * Must require therapy, as determined by progressive cytopenias or symptoms (fever, night sweats, weight loss, or fatigue)
    * Must have received ≥ 2 therapies
  * Stratum 2: Mantle cell lymphoma, as determined by the presence of cyclin D1 staining OR t(11;14)
  * Stratum 3: Intermediate grade B-cell NHL, including diffuse large B-cell NHL and T-cell rich B-cell NHL

    * Diffuse large B-cell NHL arising from an indolent NHL (i.e., transformed lymphoma) allowed
    * Ineligible for potentially curative autologous stem cell transplantation
  * Stratum 4: T-cell and natural killer-cell NHL, including anaplastic large cell lymphoma and peripheral T-cell NHL

    * Primary cutaneous lymphoma or Sezary syndrome allowed provided criteria for measurable disease are met
    * Received ≥ 1 prior systemic therapy
  * Stratum 5: Hodgkin's lymphoma

    * Any of the following subtypes are allowed:

      * Nodular sclerosing
      * Mixed cellularity
      * Lymphocyte predominant
      * Lymphocyte depleted
    * Ineligible for potentially curative autologous stem cell transplantation
  * Stratum 6: Progressive stage I or stage II or IIIA multiple myeloma meeting ≥ 1 major and 1 minor criterion OR ≥ 3 minor criteria as follows:

    * Major criteria

      * Plasmacytoma on tissue biopsy
      * Bone marrow plasmacytosis ≥ 30% of marrow cellularity
      * Monoclonal paraprotein ≥ 3,500 mg/dL (IgG), or ≥ 2,000 mg/dL (IgA), OR monoclonal protein (Bence-Jones protein) ≥ 1,000 mg by 24-hour urine collection
    * Minor criteria

      * Bone marrow plasmacytosis 10-29% of marrow cellularity
      * Monoclonal paraprotein < 3,500 mg/dL (IgG) or < 2,000 mg/dL (IgA)
      * Lytic bone lesions by x-ray or CT scan
      * Decrease in normal IgM (< 50 mg/dL), IgA (< 100 mg/dL), or IgG (< 600 mg/dL)
* Relapsed or refractory disease
* Measurable disease, defined by 1 of the following:

  * At least 1 node > 2 cm by CT scan
  * Measurable disease in a lymphoid structure (i.e., spleen) by CT scan
  * Bone marrow involvement (> 20% of marrow cellularity)
  * Patients with multiple myeloma must have detectable serum or urinary paraprotein
  * Patients with only cutaneous or subcutaneous disease (i.e., no measurable lymph node or bone marrow disease) are eligible if the extent of rash or skin involvement OR the size of the nodules are measurable
* Must have received ≥ 1 prior therapy

  * Steroids alone are not considered prior therapy for patients with NHL or Hodgkin's lymphoma
  * High-dose dexamethasone is considered 1 prior therapy for patients with multiple myeloma
* No standard effective therapy exists
* No HIV-associated lymphoma
* No nonsecretory multiple myeloma
* Performance status - ECOG (Eastern Cooperative Oncology Group) 0-2
* No concurrent hormonal therapy except steroids for new adrenal failure or hormones administered for non-disease-related conditions (e.g., insulin for diabetes)
* Hemoglobin ≥ 9.0 g/dL*
* Absolute neutrophil count ≥ 1,500/mm^3*
* Platelet count ≥ 50,000/mm^3*
* AST (aspartate aminotransferase) ≤ 3 times upper limit of normal (ULN)
* Bilirubin ≤ 2 times ULN
* No major renal dysfunction that would preclude study compliance or participation
* Phase I:

  * Creatinine ≤ 1.5 mg/dL
  * Creatinine clearance ≥ 70 mL/min
* Phase II:

  * Creatinine ≤ 2.0 mg/dL
  * Creatinine clearance ≥ 50 mL/min
* No cardiac or vascular dysfunction that would preclude central venous access, vigorous hydration, or hemodialysis
* No other major cardiac dysfunction that would preclude study compliance or participation
* No major pulmonary dysfunction that would preclude study compliance or participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No chronic gastrointestinal disease (e.g., Crohn's disease, ulcerative colitis, or short gut syndrome) that would preclude study compliance or participation
* No other major organ system (including neurological or psychiatric) dysfunction that would preclude study compliance or participation
* Prior radiotherapy, including radioimmunotherapy, allowed
* No concurrent radiotherapy
* Prior idiotype vaccination or stem cell transplantation allowed
* More than 6 weeks since prior mitomycin or nitrosoureas
* No other concurrent chemotherapy
* More than 4 weeks since other prior therapy
* Prior systemic steroids allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-12; Primary Completion 2011-02 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jones, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Hofmeister CC, Poi M, Bowers MA, Zhao W, Phelps MA, Benson DM, Kraut EH, Farag S, Efebera YA, Sexton J, Lin TS, Grever M, Byrd JC. A phase I trial of flavopiridol in relapsed multiple myeloma. Cancer Chemother Pharmacol. 2014 Feb;73(2):249-57. doi: 10.1007/s00280-013-2347-y. Epub 2013 Nov 16. PMID 24241210

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were accrued to the study between April 2006 and September 2010.
Pre-assignment Details: Patients with confirmed diagnosis of NHL (Non-Hodgkin's lymphoma) were accrued to one of the four cohorts defined by the World Health Organization criteria: indolent B-cell, mantle cell, intermediate-grade B-cell including transformed lymphoma and T-/NK-cell excluding primary cutaneous disease.
Groups:
- Dose Level 1 (Flavopiridol 30 mg/m2 + 30 mg/m2); Dose Level 2 (Flavopiridol 30 mg/m2 + 50 mg/m2); Dose Level 3 (Flavopiridol 50 mg/m2 + 50 mg/m2): Patients receive flavopiridol IV over 4½ hours on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dose Level 1 (Flavopiridol 30 mg/m2 + 30 mg/m2) | Dose Level 2 (Flavopiridol 30 mg/m2 + 50 mg/m2) | Dose Level 3 (Flavopiridol 50 mg/m2 + 50 mg/m2)
Started | 13 | 19 | 14
Patients Evaluable for Toxicity | 11 | 12 | 12
Completed | 11 | 12 | 12
Not Completed | 2 | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Alvocidib): PHASE I: Patients receive flavopiridol IV over 4½ hours on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  PHASE II: Patients receive flavopiridol* as in phase I at the MTD determined in phase I.
  alvocidib: Given IV
Arm/Group | Treatment (Alvocidib)
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 66 [34 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 26
Region of Enrollment [Number; unit: patients]
  United States | 45
  Canada | 1
Eastern Cooperative Oncology Group (ECOG) Performance status [Number; unit: patients]
  0 (Fully active) | 8
  1 (Restricted in physically strenuous activity) | 34
  2 (Ambulatory capable of all selfcare) | 4
Diagnosis [Number; unit: patients]
  Indolent B-cell | 15
  intermediate grade B-NHL | 17
  Mantle cell lymphoma | 7
  T/NK cell NHL | 7

OUTCOME MEASURES:

1. Primary Outcome: Disease-specific Dose-limiting Toxicity and Maximum Tolerated Dose of Flavopiridol Graded According to the CTCAE (Common Toxicity Criteria for Adverse Effects) Version 4.0 (Phase I)
Description: Dose limiting toxicity (DLT) for an individual disease group is defined as 1) any grade 3-4 non-hematologic toxicity (except leukopenia or neutropenia) that does not resolve or decrease to grade 1-2 within 2 weeks, or 2) any grade 4 hematologic toxicity that causes more than a 1 week delay in administration of therapy.
Time Frame: 28 days
Measure: Number; unit: patients
Groups:
- Dose Level 1 (Flavopiridol 30 mg/m2 + 30 mg/m2); Dose Level 2 (Flavopiridol 30 mg/m2 + 50 mg/m2); Dose Level 3 (Flavopiridol 50 mg/m2 + 50 mg/m2): PHASE I: Patients receive flavopiridol IV over 4½ hours on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  PHASE II: Patients receive flavopiridol* as in phase I at the MTD determined in phase I.
Arm/Group | Dose Level 1 (Flavopiridol 30 mg/m2 + 30 mg/m2) | Dose Level 2 (Flavopiridol 30 mg/m2 + 50 mg/m2) | Dose Level 3 (Flavopiridol 50 mg/m2 + 50 mg/m2)
Number analyzed (Participants) | 11 | 19 | 14
patients | 0 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The maximum tolerated dose (MTD) is defined as that dose level beneath the dose at which 2 or more of 6 patients experience DLT.
Time Frame: 28 days
Measure: Number; unit: mg/m2
Groups:
- Dose Level 1 (30+30): PHASE I: Patients receive flavopiridol IV over 4½ hours on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  PHASE II: Patients receive flavopiridol* as in phase I at the MTD determined in phase I.
  alvocidib: Given IV
- Level 2 (30+50); Level 3 (50+50): PHASE I: Patients receive flavopiridol IV over 4½ hours on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  PHASE II: Patients receive flavopiridol* as in phase I at the MTD determined in phase I.
Arm/Group | Dose Level 1 (30+30) | Level 2 (30+50) | Level 3 (50+50)
Number analyzed (Participants) | 11 | 12 | 12
mg/m2 | 60 | 80 | 100

3. Primary Outcome: Complete and Partial Response Rate (Phase II)
Description: Patients were assessed for clinical response after two , four and six cycle with laboratory studies, physical exam, and CT scans. Response was evaluated using the modified NCI-sponsored Working Group Lymphoma Response Criteria.
Time Frame: Up to 2 years
Population: Includes patients enrolled with Indolent B-cell NHL, Intermediate Grade B NHL, Mantle cell NHL and T/NK-cell NHL
Measure: Number; unit: patients
Groups:
- Dose Level 1 (Flavopiridol 30 mg/m2 + 30 mg/m2); Dose Level 2 (Flavopiridol 30 mg/m2 + 50 mg/m2); Dose Level 3 Dose (Flavopiridol 50 mg/m2 + 50 mg/m2): Patients receive flavopiridol IV over 4½ hours on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
Arm/Group | Dose Level 1 (Flavopiridol 30 mg/m2 + 30 mg/m2) | Dose Level 2 (Flavopiridol 30 mg/m2 + 50 mg/m2) | Dose Level 3 Dose (Flavopiridol 50 mg/m2 + 50 mg/m2)
Number analyzed (Participants) | 12 | 17 | 14
patients
  Complete Response | 0 | 0 | 0
  Partial Response | 2 | 2 | 2

4. Primary Outcome: Qualitative and Quantitative Toxicities in Regard to Organ Specificity
Description: The NCI Common Toxicity Criteria for Adverse Events (version 3.0) were used to define and grade toxicity for patients.
Time Frame: Up to 30 days after completion of study treatment
Population: Grade 3 and 4 toxicities.
Measure: Number; unit: percentage of patients
Groups:
- Dose Levels 1, 2, 3: Dose Level 1 (30 mg/m2 + 30 mg/m2), Dose Level 2 (30 mg/m2 + 50 mg/m2), Dose Level 3 (50 mg/m2 + 50 mg/m2)
  PHASE I: Patients receive flavopiridol IV over 4½ hours on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  PHASE II: Patients receive flavopiridol* as in phase I at the MTD determined in phase I.
  alvocidib: Given IV
Arm/Group | Dose Levels 1, 2, 3
Number analyzed (Participants) | 35
percentage of patients
  Leukopenia | 86
  Neutropenia | 23
  Infection | 20
  Diarrhea | 51
  Fatigue | 34

5. Primary Outcome: Lymphoid/Plasma Cell Malignancies
Description: Identify subsets, based on levels of response (PR and SD), of lymphoid / plasma cell malignancies that are suitable for larger phase II studies designed to further evaluate the efficacy and toxicity of flavopiridol.
Time Frame: Up to 2 years
Population: Response indicated for Indolent B-cell NHL, Mantle cell NHL and T-cell NHL
Measure: Number; unit: patients
Groups:
- Cohort 1: Patients diagnosed with Indolent B-cell NHL
- Cohort 2: Patients diagnosed with Mantle Cell NHL
- Cohort 4: Patients diagnosed with T Cell NHL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 4
Number analyzed (Participants) | 13 | 6 | 6
patients
  Partial Response | 3 | 2 | 0
  Stable Disease | 0 | 0 | 3

6. Secondary Outcome: Pharmacokinetics (Area Under the Curve; AUC) of Flavopiridol
Description: Whole blood samples were collected for pharmacokinetics analysis during the first (Day 1) and fourth (Day 22) treatments during cycle 1. Samples were collected on both occasions prior to dosing and at 0.5, 1, 3, 4.5, 6, 8 and 24 hour after the start of the bolus infusion.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose on Days 1 and 22 of Cycle 1
Population: total of 71 PK (Pharmacokinetic) profiles comprising 484 plasma concentration were determined for 45 of 46 patients following treatment
Measure: Mean (Standard Deviation); unit: hr×μM
Groups:
- All Dose Levels of Alvocidib: PHASE I: Patients receive flavopiridol IV over 4½ hours on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  PHASE II: Patients receive flavopiridol* as in phase I at the MTD determined in phase I.
  alvocidib: Given IV
Arm/Group | All Dose Levels of Alvocidib
Number analyzed (Participants) | 45
hr×μM
  Day 1 | 10.404 (5.923)
  Day 22 | 11.949 (5.109)

7. Secondary Outcome: Number of Patients Reporting Acute Infusion Toxicity (e.g., Fever, Hypotension, Tumor Pain, and Dyspnea)
Time Frame: Up to 30 days after completion of study treatment
Measure: Number; unit: patients
Groups:
- All Dose Levels of Alvocidib: PHASE I: Patients receive flavopiridol IV over 4½ hours on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  PHASE II: Patients receive flavopiridol* as in phase I at the MTD determined in phase I.
  alvocidib: Given IV
Arm/Group | All Dose Levels of Alvocidib
Number analyzed (Participants) | 35
patients | 8

8. Secondary Outcome: Induced Response in Patients Independent of p53 Mutational Status
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Population: Data not available due to studies were not conducted by collaborating laboratory Investigator
Arm/Group | Dose Level 1 (Flavopiridol 30 mg/m2 + 30 mg/m2) | Dose Level 2 (Flavopiridol 30 mg/m2 + 50 mg/m2) | Dose Level 3 (Flavopiridol 50 mg/m2 + 50 mg/m2)
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Pharmacodynamic Effects of Flavopiridol on Normal Peripheral Blood Mononuclear Cells (PBMCs).
Description: The correlation of the pharmacodynamic effects of flavopiridol on normal peripheral blood mononuclear cells (PBMCs)
Time Frame: Day 1
Population: Data not available due to studies were not conducted by collaborating laboratory Investigator
Arm/Group | Dose Level 1 (Flavopiridol 30 mg/m2 + 30 mg/m2) | Dose Level 2 (Flavopiridol 30 mg/m2 + 50 mg/m2) | Dose Level 3 (Flavopiridol 50 mg/m2 + 50 mg/m2)
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Pharmacokinetics (Cmax) of Flavopiridol
Description: as for outcome 6
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose on Days 1 and 22 of Cycle 1
Measure: Mean (Standard Deviation); unit: μM
Arm/Group | All Dose Levels of Alvocidib
Number analyzed (Participants) | 45
μM
  Day 1 | 1.954 (0.886)
  Day 22 | 2.071 (0.820)

ADVERSE EVENTS:
Time Frame: Patients were assessed for clinical response after two, four and six cycles with laboratory studies, physical exam, and CT scans.
Description: NCI Common Toxicity Criteria for Adverse Events (version 3.0) was used to define and grade toxicity.
Arm/Group | Treatment (Alvocidib)
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 34/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Alvocidib) (N=35)
Leukopenia (Investigations) | 30 (30)
Neutropenia (Investigations) | 34 (34)
Lymphopenia (Investigations) | 25 (25)
Anemia (Blood and lymphatic system disorders) | 22 (22)
Thrombocytopenia (Injury, poisoning and procedural complications) | 13 (13)
Infection (Infections and infestations) | 9 (9)
Neutropenia fever (General disorders) | 4 (4)
Increased ALT/AST (Investigations) | 12 (12)
Hyperbilirubinemia (Investigations) | 6 (6)
Nausea (Gastrointestinal disorders) | 12 (12)
Vomiting (Gastrointestinal disorders) | 10 (10)
Anorexia (Gastrointestinal disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 27 (27)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 8 (8)
Cytokine Release Syndrome (Immune system disorders) | 8 (8)
Fatigue (General disorders) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less